CLINICAL TRIAL: NCT00814203
Title: The Ohio State University COPD Registry
Brief Title: A Registry of COPD Patients to be Used for Future Studies
Status: Completed | Type: Observational
Sponsor: Philip Diaz (Other)
Responsible Party: Sponsor-Investigator, Philip Diaz, Philip Diaz M.D., Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2007H0248
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic obstructive lung disease: those with a condition

SUMMARY:
To develop a cohort of COPD participants to assist study staff in determining the most likely candidates for future studies.

DETAILED DESCRIPTION:
To develop a cohort of COPD participants for study staff to determine the most likely candidates for future studies and to develop a repository of blood from subjects with COPD for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age and older who have been diagnosed with COPD by at least one of the following:

  * clinical history-a documented history of COPD, emphysema, or chronic bronchitis;
  * pulmonary function results (defined as an FEV1/FVC less than 0.7;
  * radiographic results (high-resolution CT findings of emphysema

Exclusion Criteria:

* in ability to give informed consent
* prisoners
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
This is a registry protocol to determine factors contributing to the development of chronic obstructive lung disease.

SECONDARY OUTCOMES:
To develop a repository of blood from subjects with COPD for future studies. These studies may include evaluation of biologic markers of disease severity and progression.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Diaz, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States